CLINICAL TRIAL: NCT04434508
Title: Open Versus Laparoscopic Right Hemicolectomy With Complete Mesocolic Excision and Central Vascular Ligation for Right Colon Cancer. A Randomized Prospective Study.
Brief Title: Open Versus Laparoscopic Right Hemicolectomy for Right Colon Cancer
Acronym: CME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, gastrointestinal surgical center, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: laparoscopic hemicolectomy
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Colonic Cancer
Keywords: Colonic Cancer; laparoscopic right hemicolectomy; complete mesocolic excision
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Enrolled patients in the study were randomized to either laparoscopic or open right hemicolectomy with CME and central vascular ligation. The randomization process was performed using a closed envelope method which was withdrawn in the outpatient clinic by a nurse.
Who Masked: Participant
Masking Description: Enrolled patients in the study were randomized to either laparoscopic or open right hemicolectomy with CME and central vascular ligation. The randomization process was performed using a closed envelope method which was withdrawn in the outpatient clinic by a nurse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic right hemicolectomy with CME and central v (Active Comparator): laparoscopic right hemicolectomy with CME and central v
  Interventions: Procedure: laparoscopic right hemicolectomy with CME and central v
- open right hemicolectomy with CME and central v (Active Comparator): open right hemicolectomy with CME and central v
  Interventions: Procedure: Open right hemicolectomy with CME and central v

INTERVENTIONS:
Procedure: laparoscopic right hemicolectomy with CME and central v — laparoscopic right hemicolectomy with CME and central v
  Other Names: LHC with CME
  Arms: laparoscopic right hemicolectomy with CME and central v
Procedure: Open right hemicolectomy with CME and central v — Open right hemicolectomy with CME and central v
  Other Names: ORH with CME
  Arms: open right hemicolectomy with CME and central v

SUMMARY:
The aim of this study is to demonstrate the feasibility, surgical, and oncologic outcomes of laparoscopic right hemicolectomy with CME and CVL compared to open surgery.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate the feasibility, surgical, and oncologic outcomes of laparoscopic right hemicolectomy with CME and CVL compared to open surgery.

Enrolled patients in the study were randomized to either laparoscopic or open right hemicolectomy with CME and central vascular ligation. The randomization process was performed using a closed envelope method which was withdrawn in the outpatient clinic by a nurse.

The primary outcome was the number of lymph nodes (LNs) harvested among both groups. Secondary outcomes included operative time, blood loss, postoperative complications, and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients with right colonic cancer

Exclusion Criteria:

* Patients with distant metastasis, large tumors with extra-colonic invasion emergency presentation (bowel obstruction or perforation)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
the number of lymph nodes (LNs) harvested among both groups | 30 DAYS
  the number of lymph nodes (LNs) harvested among both groups

SECONDARY OUTCOMES:
operative time | INTRAOPERATIVE
  operative time
blood loss, | intraoperative
  blood loss,
post-operative complications | 30 days
  post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Ayman E Nakeeb, Principal Investigator — Mansoura University, Gastrointestinal Surgery Center; Mohamed E el sorogy, MD, Study Director — Mansoura University, Gastrointestinal Surgery Center
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Outside U.S and Canada, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months
Access Criteria: elnakeebayman@yahoo.com
URL: http://www.mans.edu.eg/en/

REFERENCES:
- [Background] Cho MS, Baek SJ, Hur H, Soh Min B, Baik SH, Kyu Kim N. Modified complete mesocolic excision with central vascular ligation for the treatment of right-sided colon cancer: long-term outcomes and prognostic factors. Ann Surg. 2015 Apr;261(4):708-15. doi: 10.1097/SLA.0000000000000831. PMID 25072438
- [Result] Vajda K, Horti I, Cserni G, Bori R, Sikorszki L. [Laparoscopic and open complete mesocolic excision in right-sided colon cancer compared with open and laparoscopic surgery]. Magy Seb. 2020 Mar;73(1):23-28. doi: 10.1556/1046.73.2020.1.3. Hungarian. PMID 32172577
- [Result] Dewulf M, Kalmar A, Vandenberk B, Muysoms F, Defoort B, Claeys D, Pletinckx P. Complete mesocolic excision does not increase short-term complications in laparoscopic left-sided colectomies: a comparative retrospective single-center study. Langenbecks Arch Surg. 2019 Aug;404(5):557-564. doi: 10.1007/s00423-019-01797-8. Epub 2019 Jun 26. PMID 31243573
- [Result] Emmanuel A, Haji A. Complete mesocolic excision and extended (D3) lymphadenectomy for colonic cancer: is it worth that extra effort? A review of the literature. Int J Colorectal Dis. 2016 Apr;31(4):797-804. doi: 10.1007/s00384-016-2502-0. Epub 2016 Jan 30. PMID 26833471
- See also: Mansoura university — http://www.mans.edu.eg/en/
- Available data/document: Study Protocol: Ayman El Nakeeb — http://www.mans.edu.eg/en/ — elnakeebayman@yahoo.com